CLINICAL TRIAL: NCT05077605
Title: Electrical Impedance Tomography: Effect of Extubation on Functional Residual Capacity
Brief Title: Effect of Extubation on Respiratory Function
Acronym: PULMOVISTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2020-CHITS-001; 2021-A00785-36 (Other: Id RCB)
Record Dates: First submitted 2021-10-01; First posted 2021-10-14 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Functional Residual Capacity
Keywords: Extubation; Functional residual capacity; Electrical impedance tomography; Pulmovista; Respiratory function
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Functional residual capacity (Experimental): Functional residual capacity measure during and after extubation
  Interventions: Other: Functional residual capacity measure by electrical impedance tomography

INTERVENTIONS:
Other: Functional residual capacity measure by electrical impedance tomography — Patient functional residual capacity will be measured by electrical impedance tomography before extubation and then at 0, 10, 15 and 20 min after extubation.

SUMMARY:
The extubation phase is a risky period of anesthesia management. During this step, serious complications can arise: hypoxemia, laryngospasm, pharyngeal obstruction, pneumonia… In spite of these complications, extubation and its impact on respiratory function, particularly on the Functional Residual Capacity (FRC), remains poorly studied because of the difficulty to make bedside measurements.

The PulmoVista 500 is a clinical routine which provide effective non-invasive bedside measurements. It would be interesting to evaluate the impact of extubation on respiratory function, and more specifically FRC changes during and after extubation.

This study will allow a better physiopathological knowledge and a quality improvement patient extubation management.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the variation of functional residual capacity and its distribution before and after extubation.

Patients with scheduled surgery and receiving general anesthesia with orotracheal intubation are included and the measurements will be performed in the post-interventional monitoring room (PICU). EELI data will be collected before extubation and then at T0, then T5, T10, T15 and T20 minutes. No subsequent follow-up is required.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years
* Patient in operating room for scheduled surgery
* Patient receiving general anaesthesia with orotracheal intubation
* Patient given written consent after information
* Patient covered by social security or equivalent regimen

Exclusion Criteria:

* Patient undergoing thoracic and spinal surgery, due to the presence of dressings that interfere with measurements,
* Patient who has undergone intracerebral surgery because of possible communication difficulties upon awakening,
* Patients with a body mass index (BMI) > 50 (measurements not possible)
* Pregnant or breastfeeding patient,
* Patient contraindicated to the use of a thoracic electroimpedancemetry technique: dressings, wounds, presence of a pacemaker, defibrillator or any other active implant.
* Patient deprived of liberty by a judicial or administrative decision or patient subject to a legal protection measure (guardianship, curatorship...)
* Patient in a period of exclusion from another research protocol
* Any other reason that, in the opinion of the investigator, could interfere with the evaluation of study objectives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
End Expiratory Lung Impedance (EELI) | Between 2 and 3 hours
  EELI variation before and at different timepoints after extubation: T0, T5, T10, T15 and T20 (min).

SECONDARY OUTCOMES:
Tidal volume distribution | Between 2 and 3 hours
  Percentage of tidal volume in the different regions of interest before extubation and at different timepoints after it: T0, T5, T10, T15 and T20 (min).
Tidal volume distribution depending on patient position | Between 2 and 3 hours
  Percentage of tidal volume according to patient position: supine with or without proclivity, lateral or ventral decubitus
Tidal volume distribution depending on surgery type and duration | Between 2 and 3 hours
  Percentage of tidal volume according to type and duration of surgery
Tidal volume distribution depending on ventilatory mode | Between 2 and 3 hours
  Percentage of tidal volume according to the ventilatory mode: controlled ventilation, spontaneous ventilation with inspiratory assistance, spontaneous ventilation of extubated patient with or without oxygenation device

CONTACTS AND LOCATIONS:
Overall Officials: Clarisse LEGER, Nurse, Study Director — Hôpital d'instruction des armées Sainte-Anne
Locations (1):
- Hôpital d'Instruction des Armées de Sainte Anne, Toulon, Var, France

IPD SHARING:
Plan to Share IPD: No